CLINICAL TRIAL: NCT03466476
Title: Evaluating the Efficacy of the TracPatch Wearable Technology on Patients Undergoing Total Knee Arthroplasty (TKA)
Brief Title: TracPatch in Total Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Consensus Orthopedics (Unknown)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Assistant Professor, Arthroplasty & Joint Reconstruction, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220990; 20171099 (Other: University of Miami)
Record Dates: First submitted 2018-03-08; First posted 2018-03-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Arthroplasty, Replacement, Knee; Osteoarthritis, Knee
Keywords: Wearable Technology; Total Knee Arthroplasty; Accelerometer
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients who meet enrollment criteria will be randomized to either the treatment group where they will receive their consensus tracpatch or be assigned to the control group where no wearable technology will be employed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Wearable Technology Group (Experimental): Patients in this arm will be provided with their own Consensus TracPatch wearable device postoperatively and instructed on its use for six weeks.
  Interventions: Device: Consensus TracPatch
- Current Standard of Care Group (No Intervention): Patients in this arm will not be provided with any wearable device. Participants will be evaluated as part of the study for a total of six weeks.

INTERVENTIONS:
Device: Consensus TracPatch — Consensus TracPatch will be attached to the participant's shin approximately two inches below the knee through use of an adhesive strip similar to a standard bandage for 6 weeks after total knee arthroplasty.
  Arms: Wearable Technology Group

SUMMARY:
Total Knee Arthroplasty is becoming an increasingly common operation. An important part of a successful overall patient outcome is regaining functional range of motion after surgery. Wearable devices for fitness have become increasingly common. This study seeks to utilize wearable technology to enhance the post-operative rehabilitation experience by allowing patients and surgeons to monitor patient recovery in real time. The Consensus TracPatch is a wearable device which utilizes an accelerometer, temperature sensor and step count to monitor patient recovery. This tool provides critical, real-time information that may offer a more complete source of data to understand a patient's postoperative clinical and rehabilitation course and guide physician postoperative management. The study hypothesizes that this new technology will improve patient postoperative mobility and patient-physician communication.

ELIGIBILITY:
Inclusion Criteria:

* Surgical candidate for total knee arthroplasty
* Greater than 18 years of age
* Have signed the written informed consent form
* Have consistent access to an iOS or Android device with Bluetooth capability

Exclusion Criteria:

* Unwilling or unable to provide consent
* Not fluent in the language of the informed consent form (English and Spanish)
* Prisoners
* Pregnant women
* Wards of the state
* Have previously undergone a TKA on that ipsilateral knee
* Deformities of > 10 degrees valgus or varus or flexion contractures of > 10 degrees.
* Considered by the surgeon to be a complex arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | Up to 6 weeks after surgery
  Range of motion, including flexion and extension of the knee will be measured with a goniometer in degrees.
  Measured in degrees, the patients range of motion in the operative knee will be measured before surgery and continuously by the TracPatch monitor up to six weeks post-operatively.

SECONDARY OUTCOMES:
Patient-Reported Outcome Measurement Information System (PROMIS) | Up to 6 weeks after surgery
  The PROMIS is a 10-question survey that assesses patient's overall functional status and ability to accomplish activities of daily living. It has a total score ranging from 9-55 with 9 indicating poor functional status.
Knee Injury and Osteoarthritis Outcome Score (KOOS Jr.) | Up to 6 weeks after surgery
  The KOOS Jr. is a standardized scoring system developed to rate both the knee prosthesis function and the patient's functional abilities after total knee arthroplasty. It has a total score ranging from 0-100 with 0 indicating more severe symptoms.
Visual Analogue Score | Up to 6 weeks after surgery
  A rating system from 1 - 10 developed to assess the patient's subjective rating of pain. A higher score indicates worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Hernandez, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belsi A, Papi E, McGregor AH. Impact of wearable technology on psychosocial factors of osteoarthritis management: a qualitative study. BMJ Open. 2016 Feb 3;6(2):e010064. doi: 10.1136/bmjopen-2015-010064. PMID 26842273
- [Background] Kleijn LL, van Hemert WL, Meijers WG, Kester AD, Lisowski L, Grimm B, Heyligers IC. Functional improvement after unicompartmental knee replacement: a follow-up study with a performance based knee test. Knee Surg Sports Traumatol Arthrosc. 2007 Oct;15(10):1187-93. doi: 10.1007/s00167-007-0351-7. Epub 2007 Jun 23. PMID 17589828
- [Background] Arosha Senanayake SM, Ahmed Malik O, Mohammad Iskandar P, Zaheer D. Assessing post-anterior cruciate ligament reconstruction ambulation using wireless wearable integrated sensors. J Med Eng Technol. 2013 Nov;37(8):498-510. doi: 10.3109/03091902.2013.837529. Epub 2013 Oct 14. PMID 24117351
- [Background] Kwasnicki RM, Ali R, Jordan SJ, Atallah L, Leong JJ, Jones GG, Cobb J, Yang GZ, Darzi A. A wearable mobility assessment device for total knee replacement: A longitudinal feasibility study. Int J Surg. 2015 Jun;18:14-20. doi: 10.1016/j.ijsu.2015.04.032. Epub 2015 Apr 10. PMID 25868424
- See also: Device website available to public — http://www.tracpatch.com/